CLINICAL TRIAL: NCT07127783
Title: The Role of a Postoperative Home Physical Therapy Program for the Treatment of Pelvic Pain in Patients Undergoing Endometriosis Excision
Brief Title: Physical Therapy After Endometriosis Excision
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Oregon Health and Science University (Other)
Responsible Party: Principal Investigator, Jacqueline Wong, Principal Investigator, Oregon Health and Science University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: STUDY00028168
Record Dates: First submitted 2025-08-11; First posted 2025-08-17 (Actual); Last update posted 2025-10-06 (Actual); Status verified 2025-09

CONDITIONS: Endometriosis; Surgery
Keywords: Active Recovery
MeSH Terms: conditions — Endometriosis

STUDY DESIGN:
Intervention Model Description: Participants will be randomized in a 1:1 ratio to either standard postoperative instructions or the active recovery intervention group.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Standard Postoperative Instructions (Active Comparator): Participants will receive standard postoperative recovery instructions
  Interventions: Behavioral: Standard Postoperative Instructions
- Active Recovery (Experimental): Participants will receive postoperative instructions to follow an active recovery protocol focused on increasing activity level, core strength exercises, and pelvic floor exercises focused on urinary and bowel symptoms. Exercises are to be completed twice per day for the 12 weeks following surgery.
  Interventions: Behavioral: Active Recovery

INTERVENTIONS:
Behavioral: Active Recovery — Participants will receive postoperative instructions to follow an active recovery protocol focused on increasing activity level, core strength exercises, and pelvic floor exercises focused on urinary and bowel symptoms. Exercises are to be completed twice per day for the 12 weeks following surgery.
  Arms: Active Recovery
Behavioral: Standard Postoperative Instructions — Standard of care postoperative instructions covering incision care, pain control, dietary instructions, and emergency precautions. Also includes guidelines regarding pelvic rest and lifting restrictions.
  Arms: Standard Postoperative Instructions

SUMMARY:
This is a randomized controlled pilot study comparing a home pelvic floor physical therapy program to routine post-operative care for patients undergoing endometriosis excisional surgery without hysterectomy. Quality of life and endometriosis symptoms will be compared following the recovery period.

DETAILED DESCRIPTION:
This is a randomized controlled pilot study conducted at a single institution comparing a home pelvic floor physical therapy program to routine post-operative care for patients undergoing endometriosis excisional surgery without hysterectomy. Patients will be recruited from a referral gynecological surgery group specializing in the diagnosis and treatment of pelvic pain and endometriosis. The goal is to assess the role of the active recovery program on quality of life and on pain and endometriosis symptoms.

Subjects will be randomized to routine post-operative care or to a home physical therapy program, in which they will receive written instruct ions and videos of exercises to complete immediately after surgery. The home exercise program was developed by the Department of Urogynecology in conjunction with pelvic floor physical therapists, and includes videos created by the education communications division. Quality of life, pain score, and endometriosis symptoms will be assessed at their pre-operative appointment, and at 6 and 12 weeks postoperatively.

ELIGIBILITY:
Inclusion Criteria:

* Premenopausal
* English speaking
* Undergoing endometriosis excision surgery without hysterectomy at Legacy Health with subspecialty-trained surgeons specializing in endometriosis care
* History of chronic pelvic pain (defined as >= 6 months of pain in the anatomic pelvis)
* Diagnosis of high tone pelvic floor dysfunction on examiniation
* Have access to reliable email and phone for study-related communication

Exclusion Criteria:

* Non-English speaking
* Unable to consent
* Unable to sustain 30 minutes of moderate activity at baseline
* Uses a mobility assistive device at baseline
* Chronic opioid use
* No histologic diagnosis of endometriosis on surgical pathology
* Need for additional pelvic rest (>2 weeks) postoperatively
* Pregnancy or planning to pursue pregnancy or undergo fertility treatments within 12 weeks postoperatively

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-08-28 (Actual); Primary Completion 2026-03 (Estimated); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
Short Form Survey (SF-36) | Collected immediately following surgery, 6 weeks following surgery, and 12 weeks following surgery
  The Short Form Survey (SF-36) is a 36-item survey regarding general health and pain and its impact on quality of life including physical activities, work, social activities, and emotional well-being over the last four weeks. Scores range from 0 to 100 with a higher score representing a more favorable health state.
Pelvic Floor Impact Questionnaire (PFIQ) | Collected immediately following surgery and 12 weeks following surgery
  The Pelvic Floor Impact Questionnaire (PFIQ) asks about how bladder, bowel, and pelvic symptoms affect the ability to do physical activities as well as their impact on emotional well-being over the last 3 months. Scores range from 0 to 300 with a lower score representing a lesser impact on quality of life.

SECONDARY OUTCOMES:
Pain Scores | Collected at baseline, 6 weeks following surgery, and 12 weeks following surgery.
  Pain measured using a Visual Analog Scale (VAS). This scale asks patients to rate their pelvic pain and dyspareunia over the last 4 weeks. Responses are on a scale from 0 to 10, with 10 being the worst pain.
Endometriosis Health Profile (EHP-5) | Collected at baseline, 6 weeks following surgery, and 12 weeks following surgery.
  The Endometriosis Health Profile (EHP-5) is a 5-item questionnaire asking about the perception of endometriosis symptoms on physical ability, emotional well-being, mood, social isolation, and appearance over the last four weeks. Scores range from 0 to 100 where 0 indicates the best health status.

CONTACTS AND LOCATIONS:
Overall Officials: Jacqueline Wong, Principal Investigator — Oregon Health and Science University
Locations (1):
- Oregon Health & Science University, Portland, Oregon, United States